CLINICAL TRIAL: NCT04511806
Title: Childhood Cancer Predisposition Study (CCPS)
Acronym: CCPS
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Christopher Porter, Associate Professor, Emory University
Other Study IDs: STUDY00000109; C3P-001 (Other: Consortium for Childhood Cancer Predisposition)
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Pediatric Cancer
Keywords: Cancer predisposition
MeSH Terms: conditions — Neoplasms | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — From the Primary Subjects:
  - Germline DNA (required), serial blood and stool samples (optional)
  From Parents and siblings
  - Germline DNA (required).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Subjects: Children (age 0-21) with a cancer predisposition syndromes (CPS).
  Interventions: Other: Registry
- Relatives of Children with CPS: Members of their Primary Family Unit will also be recruited for this study, including CPS-Affected Parents, Unaffected Parents and Siblings. Other adult family members (with documented or obligate CPS) are also eligible to enroll as Affected Family Members.
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — This prospective registry and biorepository will collect clinical data and specimens for research in childhood cancer predisposition.

SUMMARY:
The Childhood Cancer Predisposition Study (CCPS) is a multi-center, longitudinal, observational study that will collect clinical and biological data and specimens from children with a cancer predisposition syndromes (CPS) and their relatives.

The central hypothesis is that studying individuals at high risk for childhood cancer creates a unique opportunity for improving the understanding of carcinogenesis, tumor surveillance, early detection, and cancer prevention, which will collectively contribute to improving care and outcomes for pediatric patients with cancer and those with cancer predisposition syndromes (CPS).

DETAILED DESCRIPTION:
The CCPS is designed as a multi-center, longitudinal, observational study that will collect clinical and biological data and specimens from children with a CPS and their relatives. The investigators plan to:

1. Establish and maintain a framework for recruitment, participation, and surveillance of children with cancer predisposition syndromes (CPS) in clinical and translational research studies;
2. Define the natural history of disease in children with CPS; and
3. Evaluate the clinical impact and effectiveness of standard and emerging tumor surveillance strategies.

The study will enroll approximately 350 Children and 700 Relatives per year. The investigators plan to collect demographic and diagnostic data at enrollment. Longitudinal follow-up will be performed at least annually.

The CCPS includes the establishment of a biorepository, with a hub and spoke structure, with a central repository at Emory University/Children's Healthcare of Atlanta for prospective collection of some tissues, linked to local biorepositories at participating institutions. Information about inventory of tumor specimens already banked locally will be available in the database, along with reference to existing genomic studies of the tumor, such that investigators may identify and request such tissue or data for specific studies, subject to approval of the CCPS Scientific Committee.

ELIGIBILITY:
Inclusion Criteria:

Primary Subjects must meet all of the below criteria to be eligible for enrollment:

1. Be less than 21 years of age at the time of enrollment
2. Have a diagnosis of a specific CPS, whether they have had cancer or not

   * Based on clinical laboratory testing demonstrating a Pathogenic or Likely Pathogenic germline variant and/or
   * Based on well-established clinical diagnostic criteria and/or
   * Based on high clinical suspicion of a specific CPS with clinical laboratory testing demonstrating a variant of uncertain significance (VUS)

Affected Parents must meet all of the following criteria to be eligible for enrollment:

1. Be the biologic parent of a Primary Subject and
2. Carry a diagnosis (or obligate diagnosis) of the familial CPS

Adult Affected Siblings must meet all of the following criteria to be eligible for enrollment:

1. Be the biologic sibling of a Primary Subject and
2. Carry a diagnosis (or obligate diagnosis) of the familial CPS

Unaffected Parents and Siblings must meet all of the following criteria to be eligible for enrollment

1. Be the biologic parent or sibling of a Primary Subject and
2. Not carry a diagnosis (or obligate diagnosis) of the familial CPS

Affected Family Members must meet all of the following criteria to be eligible for enrollment:

1. Carry a diagnosis of (or obligate diagnosis of) the familial CPS. Documentation is requested but not required.

More than one child from a Primary Family Unit may be a Primary Subject. An Unaffected Sibling may be reclassified as a Primary Subject if diagnosed with a CPS during childhood.

Exclusion Criteria:

* Individuals with a strong personal or family history of cancer without a genetic or clinical diagnosis of a specific CPS are not eligible for enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Primary Subjects of this study are children (age 0-21) with a CPS. Members of their Primary Family Unit will also be recruited for this study, including CPS-Affected Parents, Unaffected Parents and Siblings. Other adult family members (with documented or obligate CPS) are also eligible to enroll as Affected Family Members.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Establish and maintain a framework for recruitment, participation, and surveillance of children with cancer predisposition syndromes (CPS) in clinical and translational research studies. | Up to 10 years
  This multicenter registry and biorepository will be developed with the purpose of studying individuals at high risk for childhood cancer to improve care and outcomes for pediatric patients with cancer and those with cancer predisposition syndromes (CPS).
Define the natural history of disease in children with CPS. | Up to 10 years
  To define the natural history of disease in children with CPS.
Evaluate the clinical impact and effectiveness of standard and emerging tumor surveillance strategies. | Up to 10 years
  Evaluate the clinical impact and effectiveness of standard and emerging tumor surveillance strategies to improve care and outcomes for pediatric patients with cancer and those with cancer predisposition syndromes (CPS).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Porter, MD, Principal Investigator — Emory University; Anita Villani, MD, Principal Investigator — The Hospital for Sick Children
Locations (7):
- United States (6):
  - Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual participant data reported in publications
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: * Researchers who provide a methodologically sound proposal, to achieve the aims in the approved proposal
  * Proposals should be directed to chris.porter@emory.edu. Requests will be reviewed by the study committee. Access to data will require a data access agreement.